CLINICAL TRIAL: NCT03000621
Title: Comparative Study of Circulating microRNA Changes in Patients With Liver Injury and Healthy Subjects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Electronic Science and Technology of China (Other)
Collaborators: Chengdu Nuoen Biotechnologies, Inc. (Other); Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Uestc500
Record Dates: First submitted 2016-12-17; First posted 2016-12-22 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2016-10

CONDITIONS: Drug-Induced Liver Injury; Liver Failure
Keywords: MicroRNA; miR-122; Diagnosis; Prognosis
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury; Liver Failure; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood extraction from subjects subsequently separated to plasma

GROUPS / COHORTS (2):
- Patients with liver injury
- Healthy subjects

SUMMARY:
The objectives are to:

1. validate a panel of tissue-specific miRNAs that are differentially expressed in the plasma of patients with and without liver injuries
2. investigate the physiological range of the circulating miRNA panel in Healthy Subjects and under stress
3. investigate the dysregulation of circulating miRNA panel and their prognostic and predictive values in clinical outcomes in identifying patients at high risk for mortality and acute liver failure.

This trial involves peripheral blood sampling from subjects at their earliest presentation and remaining stays in the hospitalization in the emergency department. The investigators will develop panels of miRNAs that are specific indicator of early onset of major organ failures, and correlate clinical outcomes with these miRNAs.

DETAILED DESCRIPTION:
The ICU patients after surgery or under chemotherapies in sponsor's institutes will be enrolled in this observational cohort of investigation. Whole blood samples will be separated immediately into plasma for storage. The participants will have their 2nd and 3rd samples obtained at 24-48 hours and 48-72 hours respectively. The schedule of most of sampling schedule is designed in concordance with the ICU routines to avoid extra burdens on patients. The plasma samples will be used as prognostic markers in prognostic and predictive values in identifying patients at high risk for mortality and acute liver failure. Patients who are discharged will be tracked for any clinical recurrence of the diseases every 28 days to assess the diagnostic accuracy of the miRNA biomarkers that are measured.

The 2nd objective will be assessed by measuring the concentration of miRNAs in recruited healthy volunteers before and after a brief public speech. The circulating miRNAs will be detected directly from 1 - 5 ul of plasma samples with the miRFLP assay. This capillary electrophoresis-based miRNA quantification method detects multiple miRNAs in absolute copy number in smaller sample signature with negligible batch to batch variation, thus providing a standardizable miRNA detection method.

ELIGIBILITY:
Inclusion criteria for healthy controls:

Adults 18 years and above

Exclusion criteria for healthy controls:

Underlying chronic inflammatory condition (e.g. inflammatory bowel disease) Underlying autoimmune disease (e.g. rheumatoid arthritis, systemic lupus erythematosus) Pre-existent liver disorder User of any prescribed medicine or over the counter drugs in prior 7 days.

Inclusion criteria for subjects:

Adults 18 years and above Has condition related to ICU enrollment cause

Exclusion criteria for subjects:

Age below 18 years Known pregnancy Treating physician deems aggressive care unsuitable Unable to provide informed consent or comply with study requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This research project will recruit a cohort of prospective observational cancer patients in ICU after surgery or chemotherapy. Admitted patients will be followed-up in the inpatient units in concordance with ICU protocols. Upon discharged, patients will be followed-up in every 28 days for any disease recurrence and clinical outcomes. Healthy controls will also be recruited to demonstrate the physiological level of different circulating miRNAs.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
The concentration of circulating miRNA expression quantitated in absolute copy numbers in ICU patients and their correlation with liver failure | Three years
  The concentration of circulating miRNAs in absolute quantification in comparison to the severity of liver injury (control vs. liver injury vs. acute liver injury). To investigate the potential prognosis of liver failure by the expression difference of the miRNA panel at the onset of liver injury. Sensitivity, specificity and the potential scopes of selected miRNA in the miRNA panel to distinguish different severity of liver injury and against standard clinical parameters, serum amonotransferases (ALT, AST), total bilirubin measurement.

SECONDARY OUTCOMES:
The possible physiological range of selected miRNAs in healthy subjects and the performance metrics of the miRNA detection methodology | Three years
  The concentration of circulating miRNAs in healthy subjects under resting condition and/or under stress. To investigate the potential physiological levels of the miRNA panel in healthy control as baselines.

CONTACTS AND LOCATIONS:
Overall Officials: Huang Jian, PhD, Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China